

# Device Protocol for CLE383-P005 / NCT04865354 Title: Clinical Comparison of Two Daily Disposable Contact Lenses

Protocol Number: CLE383-P005

Development Stage of

Project:

Product Support

Sponsor Name and

Address:

Alcon Research, LLC and its affiliates ("Alcon")

6201 South Freeway

Fort Worth, Texas 76134-2099

Test Product: PRECISION1<sup>™</sup> (verofilcon A) Soft Contact Lenses

(PRECISION1)

Property of Alcon Confidential

May not be used, divulged, published, or otherwise disclosed without the consent of Alcon

Document ID: V-CLN-0006649

Status: Approved, Version: 1.0  Approved Date: 10 Apr 2021

**Investigator Agreement:** 

• I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practice (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, all applicable regulatory authority regulations, and conditions of approval imposed by the reviewing IRB or regulatory authority.

- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current investigator's brochure, product information, or other sources provided by the sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical investigators and all other pertinent requirements of the sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you | ever been disqualified as an investigator by any | Regulatory Authority? |
|---|---|---|---|
| | □ No | □Yes | |
| | Have you | ever been involved in a study or other research | that was terminated? |
| | □ No | □Yes | |
| | If yes, plea | ase explain here: | |
| Pr | incipal Inve | stigator: | |
| | | Signature | Date |
| | ame and pro<br>sition: | fessional | |
| A | ldress: | | |

## **Table of Contents**

| De | evice Proto | ocol for CLE383-P005 | 1 |
|---|---|---|---|
| Ta | ble of Cor | ntents | 3 |
| Lis | st of Table | PS | 5 |
| Lis | st of Figur | res | 6 |
| 1 | GLOSS | ARY OF TERMS | 7 |
| 2 | LIST OF | F ACRONYMS AND ABBREVIATIONS | 12 |
| 3 | PROTO | COL SUMMARY | 14 |
| 4 | PROTO | COL AMENDMENTS | 21 |
| | 4.1 | Amendments | 21 |
| 5 | INTROI | DUCTION | |
| | 5.1 | Rationale and Background | 21 |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | 22 |
| 6 | STUDY | OBJECTIVES | 23 |
| | 6.1 | Primary Objective(s) | 23 |
| | 6.2 | Secondary Objective(s) | 23 |
| | 6.4 | Safety Objective(s) | 24 |
| 7 | INVEST | TIGATIONAL PLAN | 24 |
| | 7.1 | Study Design | 24 |
| | 7.2 | Rationale for Study Design | 25 |
| | | 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design Adaptations | |
| | 7.3 | Rationale for Duration of Treatment/Follow-Up | |
| | 7.4 | Rationale for Choice of Control Product | 26 |
| | 7.5 | Data Monitoring Committee | 26 |
| 8 | STUDY | POPULATION | 26 |
| | 8.1 | Inclusion Criteria | 26 |
| | 8.2 | Exclusion Criteria | 27 |
| | 8.3 | Rescreening of Subjects | 28 |

| 9 | TREATN | MENTS A | DMINISTERED | 29 |
|---|---|---|---|---|
| | 9.1 | Investiga | ational Product(s) | 29 |
| | 9.2 | Other M | edical Device or Medication Specified for Use During the Study. | 32 |
| | 9.3 | Treatmen | nt Assignment / Randomization | 32 |
| | 9.4 | Treatmen | nt masking | 33 |
| | 9.5 | Accounta | ability Procedures | 35 |
| | 9.6 | Changes | to concomitant medications, treatments/ procedures | 35 |
| 10 | STUDY | | URES AND ASSESSMENTS | |
| | 10.1 | Informed | d Consent and Screening | 36 |
| | 10.2 | | ion of Study Procedures and Assessments | |
| | | 10.2.1 | Demographics | |
| | | 10.2.2 | Medical History and Concomitant Medications | |
| | | 10.2.3 | Investigational Product compliance | 37 |
| | | 10.2.4 | Adverse Event Collection: Safety Assessment | 37 |
| | | 10.2.5 | Slit Lamp Biomicroscopy: Safety Assessment | 38 |
| | | 10.2.6 | Device Deficiencies: Safety Assessment | 38 |
| | 10.3 | Unsched | uled Visits | 38 |
| | 10.4 | | nued Subjects | |
| | 10 | 10.4.1 | Screen Failures | |
| | | 10.4.1 | Discontinuations | |
| | | 10.4.3 | Schedule of Procedures and Assessments for Subjects Discontin from Investigational Product | ued |
| | 10.5 | Clinical | Study Termination | |
| | | | Follow-up of subjects after study participation has ended | |
| 11 | ADVER | SE EVEN | TS AND DEVICE DEFICIENCIES | 40 |
| | 11.1 | General | Information | 40 |
| | 11.2 | Monitori | ing for Adverse Events | 42 |
| | 11.3 | Procedur | res for Recording and Reporting | 42 |
| | 11.5 | Unmaski | ing of the Study Treatment | 44 |
| | 11.6 | | Up of Subjects with Adverse Events | |
| | 11.7 | | cy in the Clinical Study | |
| 12 | | rieghand<br>A II 212 | | 45 |

| 12.1 | Subject Evaluability | 46 |
|-----------|----------------------------------------------------------|----|
| 12.2 | Analysis Sets | 46 |
| | 12.2.1 Safety Analysis Set | 46 |
| | 12.2.2 Full Analysis Set | 46 |
| | 12.2.3 Per Protocol Analysis Set | |
| 12.3 | Demographic and Baseline Characteristics | |
| 12.4 | Effectiveness Analyses | 46 |
| | 12.4.1 Analysis of Primary Effectiveness Endpoint(s) | 47 |
| | 12.4.1.1 Statistical Hypotheses | |
| | 12.4.1.2 Analysis Methods | 47 |
| 12.5 | Handling of Missing Data | 50 |
| 12.6 | Safety Analyses | |
| 12.7 | | |
| 12.7 | interim Anaryses and Reporting | |
| 12 DATA H | IANDLING AND ADMINISTRATIVE REQUIREMENTS | 50 |
| 13.1 | Subject Confidentiality | |
| 13.2 | Completion of Source Documents and Case Report Forms | |
| 13.3 | Data Review and Clarifications | |
| 13.4 | Sponsor and Monitoring Responsibilities | |
| 13.5 | Regulatory Documentation and Records Retention | 54 |
| 13.6 | Quality Assurance and Quality Control | 55 |
| 14 ETHICS | | 55 |
| | List of Tables | |
| Table 2–1 | List of Acronyms and Abbreviations Used in This Protocol | 12 |
| Table 3–1 | Schedule of Study Procedures and Assessments | 19 |
| | • | |

| Table 6–1 | Primary Objective(s) | 23 |
|-------------|----------------------------------------------|----|
| Table 6–3 | Safety Objective(s) | 24 |
| Table 9–1 | Test Product | 29 |
| Table 9–2 | Control Product | 31 |
| | List of Figures | |
| Figure 7-1 | Flowchart of Study Visits | 25 |
| Figure 11–1 | Categorization of All Adverse Events | 41 |
| Figure 11–2 | Categorization of All Serious Adverse Events | 41 |

# 1 GLOSSARY OF TERMS

| Names of test product(s) | Throughout this document, test product(s) will be referred to as PRECISION1 (or PRECISION1 soft contact lenses) |
|---|---|
| Name of Control Product(s) | Throughout this document, test product(s) will be referred to as Clariti 1-Day (or Clariti 1-Day soft contact lenses) |
| Adverse Device Effect (ADE) | Adverse event related to the use of an investigational medical device or comparator. Note: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation; any malfunction; and use error or intentional misuse of the test product or comparator. |
| Adverse Event (AE) | Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device or comparator. Note: For subjects, this definition includes events related to the investigational medical device, comparator, or the procedures involved. For users or other persons, this definition is restricted to events related to the use of investigational medical devices. Requirements for reporting Adverse Events in the study can be found in Section 11. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. <i>Note:</i> This definition includes malfunctions, use errors, and inadequacy in the information supplied by the manufacturer including labelling related to the investigational medical device or the comparator. Requirements for reporting Device Deficiencies in the study can be found in Section 11. |

| Enrolled Subject | Any subject who signs an informed consent form for participation in the study. |
|---|---|
| Interventional Clinical Trial | A research trial that prospectively assigns, whether randomly or not, human participants or groups of humans to one or more health-related interventions to evaluate the effects on health outcomes, and/or a research trial in which diagnostic or monitoring procedures beyond standard of care are conducted and generate outcomes for use in analysis of data. |
| Investigational Product | Is defined as a preventative (vaccine), a therapeutic (drug or biologic), device, diagnostic, or palliative used as a test or control product in a clinical trial, including a product with a marketing authorization when used or assembled (formulated or packaged) in a way different from the authorized form, or when used for an unauthorized indication, or when used to gain further information about the authorized form. |
| Malfunction | Failure of a medical device to meet its performance specifications or otherwise perform as intended. Performance specifications include all claims made in the labeling of the device. The intended performance of the device refers to the intended use for which the device is labeled or marketed. |
| Nonserious Adverse Event | Adverse event that does not meet the criteria for a serious adverse event. |
| Product Complaints | Any oral, electronic, or written communication that alleges deficiencies related to the identity (labeling), quality, durability, reliability, safety, effectiveness, or performance of a marketed product, including failure of the product, labeling or packaging to meet specifications, whether or not the product is related to or caused the alleged deficiency. A complaint may allege that an adverse event or medical device malfunction has occurred. |

| Randomized Subjects | Any subject who is assigned a randomized treatment. |
|---|---|
| Serious Adverse Device<br>Effect (SADE) | Adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event. |
| Serious Adverse Event (SAE) | Adverse event that led to any of the following: Death. A serious deterioration in the health of the subject users or other persons as defined by one or more of the following: a. a life-threatening illness or injury. Note: Life-threatening means that the individual was at immediate risk of death from the event as it occurred, i.e., it does not include an event which hypothetically might have caused death had it occurred in a more severe form. b. any potentially sight-threatening event or permanent impairment to a body structure or a body function including chronic diseases. |

| | c. in-patient hospitalization or prolonged hospitalization. Note: Planned hospitalization for a preexisting condition, or a procedure required by the CIP, without serious deterioration in health, is not considered a serious adverse event. In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-patient setting. Complications that occur during hospitalization are adverse events. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious. |
|---|---|
| | <ul><li>d. a medical or surgical intervention to prevent</li><li>a) or b).</li></ul> |
| | <ul> <li>e. any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use.</li> <li>Fetal distress, fetal death, or a congenital abnormality or</li> </ul> |
| | birth defect. |
| | Refer to Section 11 for additional SAEs. |
| Serious Health Threat | Signal from any adverse event or device deficiency that indicates an imminent risk of death or a serious deterioration in the health in subjects, users or other persons, and that requires prompt remedial action for other subjects, users or other persons. |


| | Note: This would include events that are of significant and unexpected nature such that they become alarming as a potential serious health hazard or possibility of multiple deaths occurring at short intervals. |
|---|---|
| Use Error | Act or omission of an act that results in a different medical device response than intended by manufacturer or expected by user. Note: This definition includes slips, lapses, and mistakes. An unexpected physiological response of the subject does not in itself constitute a use error. |

## 2 LIST OF ACRONYMS AND ABBREVIATIONS

Table 2–1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|---|---|
| ADE | Adverse device effect |
| AE | Adverse event |
| BCVA | Best corrected visual acuity |
| CFR | Code of Federal Regulations |
| CI | Confidence interval |
| CIP | Clinical Investigation Plan |
| Clariti 1-Day or | CooperVision® Clariti® 1 day |
| Clariti 1-Day | |
| contact lenses | |
| D | Diopter(s) |
| EDC | Electronic data capture |
| FAS | Full analysis set |
| FDA | US Food and Drug Administration |
| GCP | Good Clinical Practice |
| ICF | Informed consent form |
| ICH | International Council for Harmonisation of Technical Requirements |
| | for Pharmaceuticals for Human Use |
| IEC | Independent ethics committee |
| IP | Investigational product |
| IRB | Institutional review board |
| LID | Lens identification |
| logMAR | Logarithm of the minimum angle of resolution |
| N | Number |
| N/A | Not applicable |
| NI | Noninferiority |
| OD | Right eye |
| OS | Left eye |
| PRECISION1 or | PRECISION1 (verofilcon A) Soft Contact Lenses |
| PRECISION1 | |
| contact lenses | |

| Abbreviation | Definition |
|--------------|-------------------------------|
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SLE | Slit lamp examination |
| US / USA | United States of America |
| VA | Visual acuity |
| VS | Versus |

# **3 PROTOCOL SUMMARY**



| Study Design | This is a prospective, randomized, controlled, double-masked, bilateral crossover, daily wear, multicenter clinical study. Subjects will be expected to attend 3 visits. The total duration of a subject's participation in the study will be up to 22 days. Subjects will be expected to wear their study contact lenses daily for at least 10 hours per day. The day prior to visits 2 and 3, subjects will be expected to wear the study lenses for at least 16 hours. |
|---|---|
| Subject<br>population | Volunteer subjects aged 18 or over who are habitual spherical soft contact lens wearers (excluding current/previous PRECISION1, Clariti 1-Day and DAILIES TOTAL1® habitual lens wearers), have at least 3 months of contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and at least 10 hours per day. Planned number of subjects enrolled/consented: ~173 Planned number of completed subjects: 150 |
| Key inclusion criteria (See Section 8.1 for a complete list of inclusion criteria) | <ul> <li>Successful wearers of spherical soft contact lenses with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.</li> <li>subject must possess spectacles and willing to wear habitual spectacles for vision correction when study lenses are not worn, as needed.</li> <li>Willing to wear contact lenses for at least 16 hours on one of the days (day prior to each week 1 visit).</li> </ul> |
| Key exclusion criteria (See Section 8.2 for a complete list | <ul> <li>Participation of the subject in a clinical trial within the previous 15 days or currently enrolled in any clinical trial.</li> <li>Habitual PRECISION1, Clariti 1-Day, and DAILIES TOTAL1 contact lens wearers.</li> <li>Any monovision and multifocal lens wearers.</li> </ul> |


| of exclusion | | | | |
|---|---|---|---|---|
| criteria) | | | | |
| Data analysis | Planned Data Analysis | | | |
| Data analysis | Planneu Data A | Anaiysis | | |
| | To address the p | primary | objecti | ves, |
| | | es are summarized be | | |
| | | | | <b>-</b> |
| | Endpoint | Comparison | Statistical Method | _ |
| | Primary | PREGIGIONI1 | 3.51 1.00 | _ |
| | Distance VA | PRECISION1 vs | Mixed effect repeated | |
| | | Clariti 1-Day | measures | |
| | | Noninferiority | NI margin = $0.05 (logMAR)$ | |

| Associated materials | Lubrication/re-wetting drops will not be permitted. |
|---|---|
| Key words | PRECISION1, Clariti 1-Day, daily wear, visual acuity, Visual Analog Scales, Likert |

Table 3–1 Schedule of Study Procedures and Assessments

| Procedure / Assessment | Prescreening<br>(optional) | Visit 1 Screening/Baseline/ Dispense Lens 1 | Visit 2<br>Week 1 Follow-up<br>Lens 1 / Dispense<br>Lens 2 | Visit 3<br>Week 1 Follow-up<br>Lens 2 / Exit | Unscheduled<br>Visit / Early<br>Exit |
|---|---|---|---|---|---|
| | | | 8 days after Visit 1 | 8 days after<br>Visit 2 | N/A |
| Informed Consent | - | ✓ | - | - | - |
| Demographics | - | ✓ | - | - | - |
| Medical History ‡ | - | ✓ | ✓ | ✓ | ✓ |
| Concomitant Medications ‡ | - | ✓ | ✓ | ✓ | ✓ |
| Inclusion/Exclusion | - | ✓ | - | - | - |
| Habitual lens information (brand, power) | = | ✓ | - | - | - |
| VA with habitual contact lens correction (OD, OS, LogMAR distance)* | - | ✓ | - | ✓ (Exit procedure) | (✓) |
| BCVA with manifest refraction (OD, OS, logMAR distance) | - | ✓ | (✓) | (✓) | (✓) |
| Biomicroscopy | = | ✓ | ✓ | ✓ | ✓ |
| | ī | | i | i | <u> </u> |
| | ı | | ı | | |
| Randomize | | ✓ | | - | |
| Dispense (provide) study lenses | - | ✓ | ✓ | - | (✓) |
| VA (logMAR distance) with study lenses, OD, OS | - | - | <b>√</b> | ✓ | - |

| Procedure / Assessment | Prescreening<br>(optional) | Visit 1 Screening/Baseline/ Dispense Lens 1 | Visit 2<br>Week 1 Follow-up<br>Lens 1 / Dispense<br>Lens 2 | Visit 3<br>Week 1 Follow-up<br>Lens 2 / Exit | Unscheduled<br>Visit / Early<br>Exit |
|---|---|---|---|---|---|
| | | | 8 days after Visit 1 | 8 days after<br>Visit 2 | N/A |
| | 1 | 1 | | - | ı |
| | 1 | ı | • | • | 1 |
| | I | ı | | • | I |
| | I | I | • | • | I |
| | I | ı | I | | 1 |
| AF | | L | <b>■</b> | <b>-</b> | |
| AEs Device Deficiencies | - | <b>√</b> | <b>√</b> | <b>✓</b> | <b>✓</b> |
| Exit Form | - | ( <b>√</b> ) | (✓) | (✓) | ( <b>√</b> ) |

<sup>(✓)</sup> assessment performed as necessary,

<sup>\*</sup> source only

### 4 PROTOCOL AMENDMENTS

Modification of the protocol is prohibited without prior written agreement in the form of a protocol amendment. All amendments must be created by the study sponsor and must be approved by the IRB/IEC and global and regional Health Authorities, as applicable, prior to implementation except when required to mitigate immediate safety risks or when the changes involve only logistical or administrative revisions.

Amendments may necessitate that the informed consent and other study-related material be revised. If the consent form is revised, all subjects currently enrolled in the study must sign the approved, revised informed consent (re-consent), as required by the IRB/IEC.

#### 4.1 Amendments

There are no amendments. This is the first version of the protocol.

#### 5 INTRODUCTION

### 5.1 Rationale and Background

It is estimated that soft contact lenses account for over 90% of lens fits. Furthermore, it was reported that almost 32% of soft contact lenses were prescribed in a daily disposable modality. PRECISION1 is a new daily disposable silicone hydrogel contact lens with a material that combines high oxygen transmissibility with a low modulus of elasticity. PRECISION1 contact lenses are intended for the optical correction of refractive ametropia in persons with nondiseased eyes requiring subjects to wear spectacles for vision correction. The unique properties of PRECISION1 contact lenses provide precise vision, long lasting comfort and excellent handling.

## 5.2 Purpose of the Study

The purpose of this study is to evaluate the overall clinical performance of PRECISION1 contact lenses when compared to another commercially available daily disposable contact lens, Clariti 1-Day.

### 5.3 Risks and Benefits

Contact lenses may offer improved peripheral vision and the convenience of not wearing spectacles. Material properties and design characteristics of the contact lens in development are features consistent with successful contact lens wear.

PRECISION1 and Clariti 1-Day contact lenses are for daily wear use under a daily disposable wear modality; further details on any known potential risks and benefits can be found in the package insert.

PRECISION1 and Clariti 1-Day contact lenses are not intended for use with a cleaning/disinfecting solution, and the biocompatibility with lens care solutions and any associated clinical effects are unknown.

A summary of the known potential risks and benefits associated with PRECISION1 can be found in the package insert. Risks are minimized by compliance with the eligibility criteria and study procedures, and through close supervision by a licensed clinician during exposure to the study lenses.

The site personnel will educate subjects on proper hygiene and lens handling, and compliance with the use of contact lenses according to the protocol. Subjects should be instructed not to wear contact lenses while sleeping or swimming. The site personnel will also advise the subjects to remove contact lenses and return for prompt follow-up of symptoms, such as ocular discomfort, foreign body sensation, excessive tearing, vision changes, or hyperemia.

There may also be unknown risks to use of these study contact lenses. Any risk to subjects in this clinical study will be minimized by compliance with the eligibility criteria and study procedures, clinical oversight and monitoring.

## **6 STUDY OBJECTIVES**

# 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| To demonstrate noninferiority in the visual | Distance VA with study lenses (OD, OS; |
| acuity at distance when wearing | logMAR) |
| PRECISION1 contact lenses compared to | |
| Clariti 1-Day contact lenses. | |

# **6.2** Secondary Objective(s)

Not Applicable.

# **6.3** Exploratory Objective(s)





### 6.4 Safety Objective(s)

Table 6–3 Safety Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Describe the safety profile of the study | • AEs |
| products | <ul> <li>Biomicroscopy findings</li> </ul> |
| | <ul> <li>Device deficiencies</li> </ul> |

### 7 INVESTIGATIONAL PLAN

## 7.1 Study Design

This is a prospective, randomized, controlled, double-masked bilateral crossover, daily wear, multi-center clinical study. Habitual soft contact lens wearers will be randomized in 1 of the 2 crossover sequences. Subjects and investigators will be masked. An unmasked study staff member will prepare the contact lenses for dispensing.

Subjects will be expected to attend 3 visits: Screening/Baseline/Dispense Lens 1, Week 1 Follow-up Lens 1, Week 1 Follow-up Lens 2/Exit. The total duration of a subject's participation in the study will be up to 22 days. Subjects will be expected to wear their study contact lenses daily for at least 10 hours per day.

On the day prior to visits 2 and 3, subjects will be instructed to wear the study lenses at least 16 hours.

Figure 7-1 Flowchart of Study Visits



## 7.2 Rationale for Study Design

The crossover design will ensure that the same subject is exposed to both the test and control lens materials; therefore, objective assessments will be obtained for both lenses from the same subject. The study will include only those subjects who are current wearers of spherical soft contact lenses in both eyes with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.

Furthermore, the subjects will not be permitted to use lubrication/rewetting drops during the duration of the study as this may confound the primary effectiveness endpoint. The study will exclude any habitual PRECISION1, Clariti 1-Day and DAILIES TOTAL1 contact lens wearers in the past 3 months prior to consent in order to reduce potential bias of wearers to their habitual contact lenses. The study will also exclude subjects who wish to wear their contact lenses in monovision modality during the study and multifocal lens wearers.

# 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design Adaptations

An interim analysis will not be performed.

### 7.3 Rationale for Duration of Treatment/Follow-Up

Subjects will wear each study product bilaterally for approximately 1 week. The lenses will be provided by a qualified unmasked study staff member in such a manner that the subject and the investigator remain masked to the lens type. The primary variable will be assessed on approximately after 1 week of wearing each study product

### 7.4 Rationale for Choice of Control Product

Clariti 1-Day contact lenses were chosen as the control product because these lenses have the same wear modality and replacement schedule.

### 7.5 Data Monitoring Committee

Not applicable.

### 8 STUDY POPULATION

The study population consists of male and female subjects aged 18 or over who are wearers of spherical soft contact lenses in both eyes with a least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day. Subjects who are current or previous PRECISION1, Clariti 1-Day, and DAILIES TOTAL1 habitual lens wearers will be excluded

This study aims to enroll (consent) approximately 173 subjects in approximately 10 sites in the US, with a target of 150 completed subjects.

### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject is considered enrolled in the study.

Subjects eligible for inclusion in this study must fulfill **all** of the following criteria:

- 1. Subjects must be  $\geq$  18 years of age.
- 2. Subjects must be able to understand and must sign an informed consent form (ICF) that has been approved by an Institutional Review Board (IRB/IEC).

Status: Approved, Version: 1.0

Approved Date: 10 Apr 2021

3. Current wearers of any commercial spherical soft contact lenses with at least 3 months wearing experience, with a minimum wearing time of 5 days per week and 10 hours per day.



- 7. Subject must be willing to wear contact lenses for at least 16 hours of lens per day on one of the days (day prior to each week 1 visit).
- 8. Subject must possess spectacles and willing to wear habitual spectacles for vision correction when study lenses are not worn, as needed.



### 8.2 Exclusion Criteria

Subjects fulfilling any of the following criteria are not eligible for participation in this study.

1. Current/previous PRECISION1, Clariti 1-Day, and DAILIES TOTAL1 habitual lens wearers and any monovision & multifocal lens wearers.





# 8.3 Rescreening of Subjects

Rescreening of subjects is not allowed in this study.

### 9 TREATMENTS ADMINISTERED

# 9.1 Investigational Product(s)

Test Product(s): PRECISION1 soft contact lenses

Control Product(s) (If applicable): Clariti 1-Day soft contact lenses

Table 9–1 Test Product

| Test Product | PRECISION1 soft contact lenses |
|---|---|
| Manufacturer | Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, Texas 76134-2099 USA |
| Indication for use and intended purpose in the current study | Precision1 spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with nondiseased eyes with up to approximately 1.50 D of astigmatism that does not interfere with visual acuity. |
| Product description<br>and parameters<br>available for this<br>study | <ul> <li>Material: verofilcon A</li> <li>Water content: 51%</li> <li>Power range: -1.00 to -6.00 D in 0.25 D steps</li> <li>Base curve (mm): 8.3</li> <li>Diameter (mm): 14.2</li> </ul> |
| Formulation | Please see the package insert |
| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>Bilateral</li> </ul> </li> <li>Replacement period: Daily Disposable</li> <li>Exposure: <ul> <li>16 days total duration (test and control)</li> <li>Test Product: 8 days</li> <li>Control Product: 8 days</li> </ul> </li> <li>Lens Care: N/A</li> </ul> |



Table 9–2 Control Product

| Control Product(s) | Clariti 1-Day soft contact lenses |
|---|---|
| Manufacturer | Cooper Vision 711 North Road Scottsville, New York 14546 USA |
| Indication for Use | Clariti 1-Day soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with nondiseased eyes that may exhibit astigmatism up to 2.00 D that does not interfere with visual acuity. |
| Product description<br>and parameters<br>available for this<br>study | <ul> <li>Material: somofilcon A</li> <li>Water content: 56%</li> <li>Power range: -1.00 to -6.00 D in 0.25 D steps</li> <li>Base curve (mm): 8.6</li> <li>Diameter (mm): 14.1</li> </ul> |
| Formulation | Please see the package insert |
| Usage | <ul> <li>Wear: <ul> <li>Daily Wear</li> <li>Bilateral</li> </ul> </li> <li>Replacement period: Daily Disposable</li> <li>Exposure: <ul> <li>16 days total duration (test and control)</li> <li>Test Product: 8 days</li> <li>Control Product: 8 days</li> </ul> </li> <li>Lens Care: N/A</li> </ul> |



More information on the test and control products can be found in the respective Package Inserts.

# 9.2 Other Medical Device or Medication Specified for Use During the Study

No other medical devices or medications are required to be used in conjunction with the treatments during the clinical study.

## 9.3 Treatment Assignment / Randomization

Subjects will be randomized in a 1:1 ratio to receive treatment with Test product then Control product or Control product then Test product, respectively.

Only after signing the ICF, a subject will be assigned a subject number by the electronic data capture system.

Status: Approved, Version: 1.0

Approved Date: 10 Apr 2021

A randomization list will be generated using a validated system that automates the random assignment of treatments (lens sequence) to randomization numbers in the specified ratio. Subjects will be assigned treatment (lens sequence) according to the randomization list uploaded in the randomization system. The randomization list will be generated and maintained by the study sponsor.

At Visit 1, all eligible subjects will be randomized via the EDC/randomization integration system to one of the treatments (lens sequence). The investigator or delegate will access the respective system after confirming that the subject meets all the eligibility criteria. The EDC/randomization integration system will inform the site user of the treatment (lens sequence) assignment to be dispensed to the subject.

## 9.4 Treatment masking

This study is double-masked, with subjects randomized to use the PRECISION1 contact lenses and the Clariti 1-Day contact lenses for the duration 1-week treatment period, per lens type.





This level of masking will be maintained throughout the conduct of the study. Unmasking will occur only after all planned study data have been validated, and the database locked.



9.5 Accountability Procedures

It is the investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- All unused products are available for return to the study sponsor, as directed
- Any study lenses associated with a device deficiency or with any product-related adverse
  event (i.e., ADE or SADE) are returned to the study sponsor for investigation, unless
  otherwise directed by the sponsor. Refer to Section 11 of this protocol for additional
  information on the reporting of device deficiencies and AEs and the return of study
  products associated with these events.

## 9.6 Changes to concomitant medications, treatments/ procedures

After the subject is enrolled into the study, the investigator must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications,
- Any medical procedure or hospitalization that occurred or is planned
- Any nondrug therapies (including physical therapy and blood transfusions).

The investigator must document this information in the subject's case history source documents.

### 10 STUDY PROCEDURES AND ASSESSMENTS

Subjects will be expected to attend 3 office visits, as shown below.

| Visit # | Visit Type | Visit Window |
|---------|---------------------------------|----------------------|
| Visit 1 | Screen/Baseline/Dispense Lens 1 | N/A |
| Visit 2 | Week 1 Follow-up Lens 1 | 8 days after Visit 1 |
| Visit 3 | Week 1 Follow-up Lens 2/Exit | 8 days after Visit 2 |

Unscheduled Visits and Early Termination Visits are allowed, if necessary.

Study lenses will be provided to the subjects to take home for daily wear during the course of the trial.

Study randomization will occur at Visit 1 with assigned lenses provided to take home at Visit 1 and Visit 2.

Lubrication/rewetting drops will not be permitted during this study.

### 10.1 Informed Consent and Screening

The investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF BEFORE any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining
consent from the subject and a witness, if applicable, sign and date the informed consent document.

Status: Approved, Version: 1.0

Approved Date: 10 Apr 2021

The investigator or delegate must provide a copy of the signed document to the subject and place the original signed document in the subject's chart, or provide documentation as required by local regulations.

Optional prescreening for eligibility of potential subjects must be done using the using the IRB-approved script and symptomatology questionnaire.

## 10.2 Description of Study Procedures and Assessments

All study procedures and assessments are to be performed according to the table of procedures (Table 3-1). The investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

## 10.2.1 Demographics

Obtain demographic information including age, race, ethnicity, and sex.

## 10.2.2 Medical History and Concomitant Medications

| Collect medical history information, including information on all medications used with | hin the |
|---|---|
| past 30 days. | |

# 10.2.3 Investigational Product compliance

Review subject compliance with the IP usage

# 10.2.4 Adverse Event Collection: Safety Assessment

Assess and record any adverse events that are observed or reported, including those associated with changes in concomitant medication dosing since the previous visit in the subject source documents. See Section 11 for further details regarding AE collection and reporting.

# 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment

SLE of the cornea, iris/anterior chamber and lens must be performed in both eyes before instillation of any diagnostic eye drops.

## 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any device deficiencies that are reported or observed, including those associated with changes in concomitant medication dosing since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11. Device deficiencies on comparator lenses should be reported per the manufacturer's guidelines.

#### 10.3 Unscheduled Visits

If a subject visit occurs between any regularly scheduled visits, this visit must be documented as an Unscheduled Visit. During all unscheduled visits, the investigator must conduct the following procedures:

- Collect adverse event information
- Collect device deficiency information
- Record changes in medical condition or concomitant medication
- Biomicroscopy

The investigator may perform additional procedures for proper diagnosis and treatment of the subject according to Table 3-1 or at their discretion. The investigator must document this information in the subject's case history source documents.

If during an Unscheduled Visit the subject is discontinuing the IP or discontinuing from the study, the investigator must conduct Exit procedures according to Table 3-1 Schedule of Study Procedures and Assessments and Section 10.4.3, as possible.

## **10.4 Discontinued Subjects**

#### 10.4.1 Screen Failures

Subjects who were excluded from the study after signing the informed consent and prior to randomization to study product assignment and dispensing of study product.

The investigator must document the reason for screen failure in the subject's case history source documents.

Subject numbers must not be re-used.

#### 10.4.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the investigator after signing the informed consent.

Subject numbers of discontinued subjects must not be re-used.

Subjects may discontinue from study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the investigator, continued treatment poses a risk to their health.

For subjects discontinuing from the study, the investigator must complete all Exit procedures according to Table 3-1 Schedule of Study Procedures and Assessments and Section 10.4.3, if the subject is willing and able, and if in the opinion of the investigator it is safe for the subject to do so.

The investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

# 10.4.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product

Other than screen failures, if a subject discontinues from the study, the subject should undergo an Early Exit Visit. Refer to Table 3-1.

## 10.5 Clinical Study Termination

The study sponsor reserves the right to close the investigational site or terminate the study in its entirety at any time.



## 10.5.1 Follow-up of subjects after study participation has ended

Following this study, the subject will return to their eye care professional for their routine eye care.

#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

Comprehensive adverse event data will be collected in the subject source records. All AEs will be reported in the eCRF, however adverse event details collected will be determined based on the type of AE (ocular or systemic), if serious criterion is met, relationship to the IP, or if a subject discontinues due to the AE.

#### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). Refer to the Glossary of Terms for categories of AEs and SAEs.

Figure 11–1 Categorization of All Adverse Events



Figure 11–2 Categorization of All Serious Adverse Events



#### **Device Deficiencies**

A device deficiency may or may not be associated with subject harm (i.e., ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The investigator should

determine the applicable category for the identified or suspect device deficiency and report any subject harm separately.

- Event 1
- Event 2
- Event 3, etc.

## 11.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the investigator should inquire about AEs by asking the standard questions shown below and report as applicable:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take since your last study visit?"

In addition, changes in any *protocol-specific parameters* and/or *questionnaires* evaluated during the study are to be reviewed by the investigator. Any untoward (unfavorable and unintended) change in a *protocol-specific parameter* or *questionnaire response* that is clinically relevant, in the opinion of the investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

# 11.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent. Any preexisting medical conditions or signs/symptoms present in a subject prior to the start of the study (i.e., before informed consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.

For each recorded event, the ADEs and SAEs documentation must include: date of occurrence, severity, treatment (if applicable), outcome, and assessments of the seriousness and causality. In addition, the investigator must document all device deficiencies reported or observed with test and control products on the Device Deficiency eCRF. The site must submit all available information on ADEs, SAEs, and device deficiencies to the study sponsor immediately as follows:

• All SAEs must be reported immediately (within 24 hours) of the investigator's or site's awareness.

• ADEs that do not meet seriousness criteria and device deficiencies must be reported within 10 calendar days of the investigator's or site's awareness.

11.5 Unmasking of the Study Treatment Masked information on the identity of the assigned medical device should not be disclosed during the study (see Section 9.4).

Status: Approved, Version: 1.0

Approved Date: 10 Apr 2021

## 11.6 Follow-Up of Subjects with Adverse Events

The investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.



# 11.7 Pregnancy in the Clinical Study

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be included in the Medical History section of the eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study.

#### 12 ANALYSIS PLAN

Continuous variables will be summarized using the number of observations, mean, standard deviation (SD), median, minimum, and maximum, as well as confidence intervals (CIs) or confidence limits where applicable. Categorical variables will be summarized with frequencies and percentages from each category.

Any deviations to the analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

## 12.1 Subject Evaluability

Final subject evaluability must be determined prior to breaking the code for masked treatment (lens sequence) assignment and locking the database, based upon the Deviations and Evaluability Plan (DEP).

## 12.2 Analysis Sets

## 12.2.1 Safety Analysis Set



## 12.2.2 Full Analysis Set

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study lenses evaluated in this study.

# 12.3 Demographic and Baseline Characteristics

Demographic information will be summarized by lens sequence and overall. Frequencies and percentages will be presented for categorical variables such as sex, age group, race, and ethnicity. Number of observations, mean, SD, median, minimum, and maximum will be presented for continuous variables such as age

# 12.4 Effectiveness Analyses



## 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary objective of this study is to demonstrate noninferiority in distance VA when wearing PRECISION1 contact lenses compared to Clariti 1-Day contact lenses. The primary endpoint is distance VA with study lenses, collected for each eye in logMAR.

## 12.4.1.1 Statistical Hypotheses

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.05 for noninferiority:

H<sub>0</sub>: 
$$\mu_{(T)} - \mu_{(C)} \ge 0.05$$
  
H<sub>a</sub>:  $\mu_{(T)} - \mu_{(C)} \le 0.05$ 

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the mean distance VA for PRECISION1 and Clariti 1-Day, respectively, on the logMAR scale.

## 12.4.1.2 Analysis Methods

A mixed effect repeated measures model will be utilized to test these hypotheses. The model will include terms for lens, visit, lens by visit interaction, period, and sequence. Withinsubject correlation due to eye and the crossover design will also be accounted for in the model. Lens difference (PRECISION1 minus Clariti 1-Day) and the corresponding one-sided 95% upper confidence limit will be computed. Noninferiority in distance VA will be declared if upper confidence limit is less than 0.05.







## 12.5 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out for the primary and key exploratory effectiveness analyses.

# 12.6 Safety Analyses

The safety endpoints are:

- AEs
- Biomicroscopy findings
- Device Deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters.

All AEs occurring from the time a subject signs informed consent to study exit will be accounted for in the reporting. Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. Descriptive summaries (frequencies and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities

Preferred Terms. AEs leading to study discontinuation, significant nonserious AEs, and SAEs will be identified. Individual subject listings will be provided, as necessary.



No inferential testing will be conducted for the safety analyses.

## 12.7 Interim Analyses and Reporting

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.



Approved Date: 10 Apr 2021

Status: Approved, Version: 1.0

# 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

# 13.1 Subject Confidentiality

| The investigator must ensure that the subject's anonymity is maintained throughout the |
|---|
| course of the study. |



# 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the study sponsor and are independent of study site staff.

If electronic records are maintained, the method of verification must be determined in advance of starting the study.





#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

## 13.4 Sponsor and Monitoring Responsibilities

The study sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and well-being of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.



# 13.5 Regulatory Documentation and Records Retention

The investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the study sponsor and the investigator's files will be reviewed as part of the ongoing study monitoring. Financial information is to be kept separately.



#### 14 ETHICS



The investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements and/or GCP must be recorded and reported to the sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records. Use of waivers to deviate from the clinical protocol is prohibited.



The study sponsor assures that the key design elements of this protocol will be registered on www.clinicaltrials.gov as required by current regulations and, if applicable, other public databases as required by local country regulations. In addition, results of this study will be made publicly available on www.clinicaltrials.gov regardless of outcome as required by current regulations and, if applicable, in other public databases as required by local country regulations.



Signature Page for V-CLN-0006649 v1.0

